CLINICAL TRIAL: NCT06110715
Title: Quantifying tACS-driven Improvement of Working Memory in Depression
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no participants enrolled
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: PSYCH-2023-31635
Record Dates: First submitted 2023-10-16; First posted 2023-11-01 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Sham Comparator): participants with depressive disorder
  Interventions: Other: sham tACS stimulation
- Active group (Experimental): participants with depressive disorder
  Interventions: Other: theta tACS stimulation

INTERVENTIONS:
Other: theta tACS stimulation — The low intensity transcranial electrical stimulation will be administered with a battery-powered, current-controlled, multi-channel stimulator from Neuroelectrics® Starstim 8. This device comes with a neoprene headcap to hold the electrodes in place. TACS will be delivered concurrently with the task. The multichannel, current-driven stimulator (Neuroelectrics StarStim 8) will be used to control independent stimulation electrodes on the scalp of the volunteer. The stimulation intensity will be up to 2 mA.
  Arms: Active group
Other: sham tACS stimulation — A placebo control stimulation will use an identical montage to the stimulation montage. However, polarities of the electrodes will be such that only a minimal amount of current reaches the brain, which is achieved through controlled current shunting between neighboring electrodes. This so-called ActiSham protocol is a verified method to imitate the sensations of actual tACS, with minimal stimulation of the brain .
  Arms: control group

SUMMARY:
TACS is an emergent method of non-invasive neuromodulation which can engage frequency-specific brain oscillations. It is increasingly recognized that neural oscillations play a system-organizing role in the brain. Evidence suggests that disorganized neural oscillations may also influence functionality of cognitive processes such as working memory. Thus, as TACS can affect neural oscillatory activity in the human brain in a non-invasive manner, it has promise to transform mental health care. The premise of this proposed work is that tACS concurrent with multi-session working memory (WM) focused skills will facilitate durable working memory and stabilized neural oscillations. Depression offers an excellent model to study the effects of tACS. The study seeka to administer 2mA of tACS using theta oscillations to improve working memory concerns associated with depression. The purpose of this study is to investigate the electrophysiological and behavioral effects of transcranial alternating current stimulation (tACS) in humans and to explore specific improvements in working memory and depressive symptoms. This study is placebo-controlled study. Participants will undergo pre- and post-assessments and either theta or sham tACS for 5 days. During each session, the volunteer will perform cognitive tasks while receiving tACS. Assessment sessions will include cognitive tasks, questionnaires, a clinical interview, and EEG.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years old.
* Stated willingness to participate and comply with all study procedures.
* Stated availability for the duration of the study.
* Meet criteria for Major Depressive Disorder.
* Agreement to adhere to lifestyle considerations throughout study duration.
* No conflict of interest with the Department of Biomedical Engineering at the University of Minnesota.
* Confident level of English language.

Exclusion Criteria:

* History or evidence of chronic neurological disorder (e.g., history of seizures, epilepsy, unexplained episodes of loss of consciousness, serious brain injury, severe or frequent headaches)
* Metal or electric implant in the head, neck or chest area.
* Implanted pacemakers or other electrically, magnetically, ir mechanically activated implant
* Vascular clips or other electrically sensitive support systems in the brain
* Serious health conditions (e.g., congestive heart failure pulmonary obstructive chronic disease, active neoplasia)
* History of head injuries.
* Pregnancy or breast-feeding.
* Significant damage of skin at sites of stimulation or other skin concerns, such as dermatitis, psoriasis, or eczema
* Alcohol or drug addiction.
* Any legal reason why the candidate cannot participate.
* Concurrent enrollment in another scientific or clinical study.
* Estimated IQ is below 70, defined by the WTAR.
* Active suicidality or other non-controlled neuropsychiatric illness. Active suicidality will be excluded based on a C-SSRS score of 3 or above in the last 6 months. Severe depression is defined as a PHQ-9 score above 20, which will also be excluded.
* A lifetime suicide attempt.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-09-05 (Actual); Primary Completion 2024-08-16 (Actual); Study Completion 2024-08-16 (Actual)

PRIMARY OUTCOMES:
working memory skills | Day 5
  Using a cognitive task that will consist of test responses (correct / incorrect) and reaction time (in ms). The task will include looking at faces expressing different emotions and matching them with previous images.
Resting state EEG | Day 6
  examine theta power and connectivity with the EEG recordings
Resting state EEG | Day 35
  examine theta power and connectivity with the EEG recordings
task-based EEG | Day 6
  examine theta power and connectivity with the EEG recordings
task-based EEG | Day 35
  examine theta power and connectivity with the EEG recordings

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Opitz, PhD, Principal Investigator — University of Minnesota; Kelvin Lim, MD, Principal Investigator — University of Minnesota